CLINICAL TRIAL: NCT01695694
Title: HIV Risk Reduction for Women Reporting Intimate Partner Violence
Brief Title: Violence and HIV Risk Among Women
Acronym: VHRW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RSRB00040309; 7K01MH080660 (NIH)
Record Dates: First submitted 2012-07-20; First posted 2012-09-28 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: HIV Risk Reduction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- community support group (Active Comparator)
  Interventions: Behavioral: community support group
- supporting positive and healthy relationships (Experimental)
  Interventions: Behavioral: supporting positive and healthy relationships

INTERVENTIONS:
Behavioral: supporting positive and healthy relationships
  Arms: supporting positive and healthy relationships
Behavioral: community support group
  Arms: community support group

SUMMARY:
The purpose of the study is to test the feasibility, acceptability, and efficacy of an adapted intervention that is theoretically and empirically guided by the Information-Motivation-Behavioral skills model (IMB) and aims at reducing sexual risk behavior among women who have experienced Intimate Partner Violence (IPV), as well as such an intervention.

DETAILED DESCRIPTION:
The two foremost health problems impacting young adult women are STDs/HIV infection and intimate partner violence (IPV). STDs pose a significant public health issue in the US, particularly among women. The consequences of some STDs are more severe for women, and include infertility, pelvic inflammatory disease, and brain, cardiovascular, and organ damage. Women with STDs are at increased risk for HIV. The proportion of AIDS cases among US adult and adolescent women has more than tripled since 1985. Approximately 12,000 US women are infected with HIV annually, primarily through heterosexual contact. Also, in the US HIV is particularly affecting women of color and those in low-income urban areas.

IPV also affects many women. While the causal links between IPV and HIV risk or infection have not yet been established, emerging empirical evidence has drawn connections between IPV with HIV risk. Several researchers have highlighted the importance of developing sexual risk reduction interventions that address the growing concern of gender-based violence against women. Also, scholars are calling for HIV prevention programs aimed at women to be more comprehensive; for example, by combining them with STD screening or with programs designed to reduce violence against women. Despite this call, there are very few empirically tested interventions for prevention and treatment targeting women who are at risk for STDs/HIV and experience IPV in their intimate relationships. To address high risk sexual behaviors among women who experience gender-based violence in their intimate relationships, I have adapted an existing information-motivation-behavioral skills (IMB) STD/HIV prevention intervention for reducing high sexual risk-taking behaviors. The STD/HIV and IPV comprehensive intervention will address both sexual risk reduction and IPV risk; the intention is to help women to acquire knowledge, skills, and strategies that will reduce their risk for both STDs/HIV and IPV.

Aim 1: To assess the feasibility and acceptability of the adapted IMB STD/HIV prevention intervention by implementing the intervention with a sample of women who are at risk for HIV/STDs and experience IPV. To achieve this aim:

1. 120 women who are at risk for HIV/STDs and have experienced IPV will be randomized either to receive the experimental prevention intervention or to attend a structurally similar drop-in enhanced support group at a domestic violence agency.
2. Enrollment, attendance, and attrition data will be used to determine the feasibility of the intervention.
3. The acceptability of the intervention will be appraised by analyzing pre- and post-intervention acceptability ratings completed by subjects and interventionists.

Aim 2: To gather preliminary evidence of the efficacy of the theoretically guided intervention using a controlled design. To achieve this aim:

1. Women in the experimental and control groups will be assessed at baseline, post-intervention, and at a 3-month follow-up.
2. Outcome analyses to calculate effect sizes for use in future power analyses for a larger RCT of the proposed intervention will include measures on primary variables of hypothesized risk antecedents, standard measures of protected and unprotected sex, and secondary variables such as mental health, self esteem, and IPV experiences.

ELIGIBILITY:
Inclusion Criteria:

Women will be eligible to participate in the research study if they meet the following criteria:

* between ages 18 and 49;
* heterosexually active;
* have experienced intimate partner violence in the last three months;
* have engaged in risky sexual behavior in the past three months;
* not currently pregnant or trying to become pregnant; and
* physically and psychologically capable of providing informed consent. All subjects will be required to provide written informed consent prior to enrolling in the study.

Exclusion Criteria:

Persons who meet one or more of the following criteria will be excluded from the study:

* men;
* women who have active psychosis or impaired mental status (confirmed with a Mini-Mental Status Exam);
* are unable to understand spoken English;
* are less than 18 years old or greater than 49 years old;
* are currently pregnant or trying to become pregnant
* women who are exclusively in same-sex relationships.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in sexual risk behavior at 3 months | at the completion of 3 months after the intervention
  Sexual risk behavior is assessed by self-reported number sexual partners in the last three months and number of episodes of unprotected sex with each partner

SECONDARY OUTCOMES:
Change from Baseline in experience of violence at 3 months | At the end 3-months after the end of the intervention
  Participant's experiences of violence as well as the frequency and intensity of thse experiences will be assessed using established measures of intimate partner violence

CONTACTS AND LOCATIONS:
Overall Officials: Mona Mittal, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States